CLINICAL TRIAL: NCT05827445
Title: Cutaneous Sensory Block Area of the Laparoscopic Assisted Transversus Abdominis Plane
Brief Title: Cutaneous Sensory Block Area of the Laparoscopic Assisted Transversus Abdominis Plane Block
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSBA-LTAP
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2022-10

CONDITIONS: Cholecystolithiasis
Keywords: Transversus abdominis plane block
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the size and location of cutaneous sensory block area after dual laparoscopic assisted transverse abdominis plane block (L-TAP) with ropivacaine in patients undergoing laparoscopic cholecystectomy.

L-TAP is applied as a medial subcostal infiltration between midclavicular and central sternal lines and a lateral subcostal infiltration between midclavicular and anterior axillary line bilaterally.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective laparoscopic cholecystectomy in a day surgery setting
* able to give oral and written consent

Exclusion Criteria:

* prior surgery to the upper abdominal wall
* known sensory deficits of the abdominal wall or thorax
* allergy to local anesthetics
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic cholecystectomy in a day surgery setting for cholecystolithiasis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cutaneous Sensory Block Area (CSBA) | 1.5 hours postoperatively
  Assessment of the CSBA was done within the duration of the cutaneous sensory effect of the laparoscopic transverse abdominis plane block. A gauze dipped in alcohol was tapped on the skin of the abdominal wall from the midsagittal line using a star-shaped approach with its center at the umbilicus to indicate cutaneous sensory changes in cold perception. Changes were marked on the skin, confirmed twice, and a connecting line drawn to determine the CSBA. The was size of the CSBA was calculated, and the location (supraumbilical or infraumbilical and medially or laterally to a vertical line through the anterior superior iliac spine.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital - North Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salmonsen CB, Lange KHW, Rothe C, Kleif J, Bertelsen CA. Cutaneous sensory block area of the laparoscopic-assisted transversus abdominis plane block. Dan Med J. 2024 Sep 9;71(10):A02240142. doi: 10.61409/A02240142. PMID 39323259